CLINICAL TRIAL: NCT00202982
Title: A Multi-Center, Randomized, Double-Blind, Parallel Group Study to Evaluate the Efficacy, Tolerability and Safety of 40 mg of Copaxone in the Treatment of Relapsing-Remitting Multiple Sclerosis Patients
Brief Title: A Study to Test the Effectiveness and Safety of a New Higher 40mg Dose of Copaxone® Compared to Copaxone® 20mg, the Currently Approved Dose
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: J. Michael Nicholas, Ph.D., Teva Neuroscience
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9006
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Relapse-Remitting Multiple Sclerosis
MeSH Terms: interventions — Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- glatiramer acetate 20 mg (Active Comparator): glatiramer acetate 20 mg
  Interventions: Drug: glatiramer acetate 20 mg
- glatiramer acetate 40 mg (Active Comparator): glatiramer acetate 40 mg
  Interventions: Drug: glatiramer acetate 40 mg

INTERVENTIONS:
Drug: glatiramer acetate 20 mg — glatiramer acetate 20 mg
  Arms: glatiramer acetate 20 mg
Drug: glatiramer acetate 40 mg — glatiramer acetate 40 mg
  Arms: glatiramer acetate 40 mg

SUMMARY:
This is a study to test if a new higher dose of Copaxone is more effective in treating relapsing-remitting multiple sclerosis than the currently available 20 mg dose.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically definite MS with disease duration (from onset) of at least 6 months.
2. Subjects must have had at least 1 documented relapse within the last year prior to study entry.
3. Subjects must have at least 1 and not more than 15 gadolinium (Gd)-enhancing lesions on the screening MRI scan.
4. Subjects must be relapse-free and not have taken corticosteroids (IV, IM and/or PO) within the 30 days prior to the screening visit.
5. Subjects must not have taken corticosteroids (IV, IM and/or PO) between the screening and baseline visits.
6. Subjects may be male or female. Women of child- bearing potential must practice a medically acceptable method of birth control. Acceptable methods include oral contraceptive, contraceptive patch, or double-barrier method (condom or IUD with spermicide).
7. Subjects must be between the ages of 18 and 50 years inclusive.
8. Subjects must be ambulatory, with a Kurtzke EDSS score of between 0 and 5 inclusive.
9. Subjects must be willing and able to give written informed consent prior to entering the study.

Exclusion Criteria:

1. Previous use of glatiramer acetate (oral or injectable).
2. Previous use of cladribine.
3. Previous use of immunosuppressive agents in the last 6 months.
4. Use of experimental or investigational drugs, including I.V. immunoglobulin, and/or participation in an investigational drug study within 6 months prior to study entry.
5. Use of interferon agents within 60 days prior to the screening visit.
6. Chronic corticosteroid (IV, IM and/or PO) treatment (more than 30 consecutive days) in the 6 months prior to study entry.
7. Previous total body irradiation or total lymphoid irradiation (TLI).
8. Pregnancy or breast feeding.
9. Patients who experience a relapse between the screening (month -1) and baseline (month 0) visits.
10. Any condition which the investigator feels may interfere with participation in the study, including alcohol and/or drug abuse.
11. A known history of sensitivity to mannitol.
12. A known sensitivity to gadolinium.
13. Inability to successfully undergo MRI scanning.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2003-08; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
The total number of T1 Gd-enhancing lesions in T1-weighted images, as measured at months 7, 8 and 9

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Cohen, MD, Study Chair — The Cleveland Clinic
Locations (20):
- United States (20):
  - Center for Neurologic Study, La Jolla, California
  - North County Neurology Associates, Oceanside, California
  - The MS Center of Atlanta, Atlanta, Georgia
  - Consultants in Neurology, Ltd, Northbrook, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - The Maryland Center for M.S., Baltimore, Maryland
  - Michigan Institute of Neurological Disorders, Farmington Hills, Michigan
  - The Minneapolis Clinic of Neurology, LTD, Golden Valley, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Clinical & Magnetic Resonance Research Ctr., Albuquerque, New Mexico
  - MSSM - Corinne Goldsmith Dickinson Center for MS, New York, New York
  - University of Rochester, Rochester, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Allegheny Neurological Associates, Pittsburgh, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
  - VAMC, Salt Lake City, Utah
  - MS Hub Medical Group, Seattle, Washington
  - Neurology & Neurosurgery, Tacoma, Washington